CLINICAL TRIAL: NCT00142402
Title: Modafinil for Improving New Learning and Memory in Multiple Sclerosis
Brief Title: Modafinil in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ndcnmss2004; PP0911
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Memory; New Learning; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
Deficits in new learning and memory in MS are a major complaint of patients, and have been noted to be a significant contributor to disability by numerous researchers. Modafinil is a psychostimulant medication, FDA approved for the treatment of Narcolepsy, with potential application for the treatment of learning and memory dysfunction in MS. This randomized clinical trial tests the efficacy of Modafinil for the treatment of new learning and memory deficits in MS.

Twenty subjects with clinically definite MS and objectively documented new learning impairment will be included in the study. All subjects will undergo baseline neuropsychological testing and EDSS to document current levels of functioning in new learning and memory abilities. Subjects will then be randomly assigned to either group 1 or group 2. Group 1 (n=10) will first undergo treatment with Modafinil (200 mg once per day in the morning) for 2 weeks. They will then undergo follow-up neuropsychological assessment and follow-up EDSS to evaluate any medication effects. After the follow-up evaluation, there will be a washout period of one week in which no medication will be administered. Group 1 will then receive a placebo medication for 2 weeks. A second follow-up evaluation will be conducted following this latter arm of the study. Group 2 (n=10) will follow the same pattern, but will receive the placebo medication during the first arm of the study and Modafinil during the 2nd arm of the study. The subjects and the experimenter administering the neuropsychological evaluation will be blind to group membership.

DETAILED DESCRIPTION:
Recent prevalence estimates of cognitive dysfunction in MS fall as high as 54-65%,21 with impairments having been documented in cognitive realms such as attention, executive control, working memory, and episodic memory. Deficits in long-term episodic memory in MS are a major complaint of patients, and have been noted to be a significant contributor to disability by numerous researchers.4,15,18 While the early studies of memory functioning in MS suggested that the memory impairment was due to difficulties in the retrieval of information from long term storage,19,26 more recent studies have challenged these conclusions. Specifically, research at KMRREC has clearly shown that verbal memory impairment in MS is primarily a function of poor acquisition of information, rather than retrieval failure.6,7,8 MS subjects require more trials to learn the same amount of information as healthy control subjects. However, once this learning has occurred, both MS and healthy control groups have comparable recall at 30-minutes, 90-minutes, and 1-week time periods (Appendix B).6,7,8 Given the apparent deficit in the acquisition of new information and the impact this deficit has on an individual's quality of life, the amelioration of this deficit is critical. The treatment of memory deficits has been the focus of research in numerous neurological populations, yet it has received little attention in MS.17 Although multiple authors have highlighted the need for cognitive rehabilitation techniques in MS,24,16 only a few existing cognitive rehabilitation programs have been aimed at improving attentional deficits,23 communication skills, 13 or memory and new learning within MS.1,2,14 In addition, few studies have examined the use of cognitive enhancing medications to treat cognitive deficits in MS. Greene and colleagues (2000) conducted a 12-week trial of Donepezil for the treatment of cognitive symptoms in MS, noting the medication to be useful for this population. Yet few other medication trials have been accomplished. Modafinil is a psychostimulant medication, FDA approved for the treatment of Narcolepsy, with potential application for the treatment of learning and memory dysfunction in MS.

Two subtypes of the glutamate receptor channels have been implicated in memory functioning, the N-methyl-D-aspartate (NMDA) and AMPA subtypes. In addition, facilitation of glutamatergic transmission has been shown to promote long-term potentiation, which is hypothesized to be involved in the encoding of new memories (e.g. 3,5). One might therefore expect improvements in new learning and memory formation with the manipulation of glutamate and aspartate receptors. In contrast, facilitation of GABA transmission induces amnesia, while inhibiting GABA transmission enhances information retention. Therefore, the inhibition of GABA should additionally enhance new learning and memory functioning. Modafinil accomplishes both of these neurochemical effects.

Animal studies have indicated that Modafinil significantly increases both aspartate and glutamate at the regional level, while decreasing the level of GABA through the inhibition of its release.20,12,10,22 In addition, Modafinil has been shown to exert its effect on specific brain regions, most notably for this study, in subregions of the hippocampus.11 Therefore, the application of Modafinil to an MS population with impairments in new learning has the potential to significantly improve cognitive functioning in this population, secondarily improving emotional symptoms and quality of life.

Modafinil has been shown to be quite safe. Headaches are the most common side effect,29,9 with other more common side effects including nausea, vomiting, nervousness, and anxiety.9 Less common, but more serious side effects have included delusions and hallucinations, palpitations, chest pain, dyspnea, increased blood pressure, and EKG changes. 9 Modafinil has been applied to the treatment of Attention Deficit Hyperactivity Disorder, with results indicating Modafinil to be a viable treatment alternative to Dextroamphetamine in ADHD,28 and TBI,9 for the treatment of underarousal. Modafinil therefore demonstrates efficacy within other patient groups with neurological impairment.

Rammohan et al 25 noted that 200mg/day of Modafinil significantly improved symptoms of fatigue in an MS sample and was tolerated quite well.25 Given that Modafinil has been proven to be a safe, effective treatment of arousal and fatigue, and its neurochemical effects are likely to enhance cognition, we are seeking to apply this medication for the treatment of cognitive deficits in MS. Due to the fact that Modafinil has been shown to act on glutamate and aspartate receptors, specifically influencing the hippocampus, it is hypothesized that treatment with this medication will result in better performance in tests of new learning and memory in an MS sample.

Participants: Twenty subjects with clinically definite MS and objectively documented new learning impairment will be included in the study. Subjects will be excluded from participation in the presence of significant language comprehension deficits. Additional exclusion criteria are as follows: age greater than 60, less than 1-month post most recent exacerbation, current treatment with corticosteroids, significant neurological history aside from MS (e.g. epilepsy, TBI), significant substance abuse history as documented by the MAST,27 significant psychiatric history (e.g. Schizophrenia, Bipolar Disorder, Major Depression), non-fluency in the English language.

Procedure: Please see study overview in Appendix C. Subjects will be recruited through physician referrals from the MS Clinic at UMDNJ in Newark, NJ (see letter of support, Appendix D). All potential subjects will undergo initial neuropsychological (NP) testing (Appendix E) to screen for study inclusion criteria, namely the presence of new learning impairment. Subjects will only be enrolled in the current protocol if they are classified as impaired in new learning and memory ability, with intact language abilities. Such impairment will be defined as performance at least 1.5 standard deviations (SD) below the mean of a healthy control sample on the Open Trial Selective Reminding Test. This test has been shown to be sensitive to deficits in new learning abilities commonly observed in MS. In addition, performance on the Token Test (see Appendix D) must be within normal limits. All subjects qualifying for the study will then undergo baseline neuropsychological testing to document current levels of functioning in new learning and memory abilities. Subjects will then be randomly assigned to either group 1 or group 2. A two-period crossover design will be used in which subjects will be randomly assigned to one of the two groups. Subjects in both groups will be seen by a physician (Dr. Greenwald) who will assess their current neurological status and complete the EDSS. Group 1 (n=10) will first undergo treatment with Modafinil (200 mg once per day in the morning) for 2 weeks. They will then undergo follow-up neuropsychological assessment and follow-up EDSS to evaluate any medication effects. After the follow-up evaluation, there will be a washout period of one week in which no medication will be administered. Group 1 will then receive a placebo medication for 2 weeks. A second follow-up evaluation will be conducted following this latter arm of the study. Group 2 (n=10) will follow the same pattern, but will receive the placebo medication during the first arm of the study and Modafinil during the 2nd arm of the study. Importantly, the subjects and the experimenter administering the neuropsychological evaluation will be blind to group membership. All subjects will be asked to keep a precise journal during both arms of the study, recording the time at which the medication was taken, any side effects, activities during the day, and any changes in cognition for each activity. They will be encouraged to contact the prescribing physician if they encounter any difficulties. See Table 1 for study protocol. A power analysis is presented in Appendix F.

Statistical Analyses: A 2 (group) x 3 (testing sessions: baseline, 15 days, 37 days) repeated measures ANOVA will be performed. We hypothesize that there will be a significant interaction of time of testing by group. Cognitive performance is expected to improve from the 1st to the 2nd testing sessions in the group 1, with just a mild practice effect documented in the group 2. Additionally, we expect a return to baseline cognitive functioning from the 2nd to the 3rd NP assessment in Group 1, with an improvement in performance noted in group 2 due to medication effects. No main effects are anticipated. A linear regression will be used to examine the influence of memory performance and perception of memory abilities on changes in depression and anxiety at the various assessment intervals. We hypothesize that as memory improves, depression and anxiety levels will decrease. Additionally, as the perception of memory improves, depression and anxiety will also decrease.

ELIGIBILITY:
Inclusion Criteria:

* Must understand English, diagnosis of Multiple Sclerosis

Exclusion Criteria:

* Significant language comprehension deficits, age greater than 60, less than 1-month post most recent exacerbation, current treatment with corticosteroids, significant neurological history aside from MS (e.g. epilepsy, TBI), significant substance abuse history as documented by the MAST,27 significant psychiatric history (e.g. Schizophrenia, Bipolar Disorder, Major Depression), non-fluency in the English language.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2003-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Scores on memory tests at 3 weeks and 6 weeks

SECONDARY OUTCOMES:
Scores on fatigue measures at 3 weeks and 6 weeks
Scores on emotional measures at 3 weeks and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D Chiaravalloti, PhD, Principal Investigator — KMRREC
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States